CLINICAL TRIAL: NCT00624910
Title: A Phase II, Single-dose, Blinded, Prospective Study to Investigate the Efficacy and Safety of the CollaRx® Bupivacaine Implant in Women Following Abdominal Hysterectomy or Other Nonlaparoscopic Benign Gynecological Procedure
Brief Title: Efficacy and Safety of a Collagen Bupivacaine Implant in Women Following Abdominal Hysterectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innocoll (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INN-CB-002
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Postoperative Pain
Keywords: Post Operative Pain; Hysterectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): A total of three 5 × 5-cm bupivacaine sponges implanted at specified layers in the wound prior to wound closure
  Interventions: Drug: Bupivacaine Collagen Sponge (CollaRx®)
- 2 (Placebo Comparator): A total of three 5 × 5-cm collagen sponges implanted at specified layers in the wound prior to wound closure
  Interventions: Drug: placebo
- 3 (No Intervention): The patient will recieve the standard of care, but no implant during surgery

INTERVENTIONS:
Drug: Bupivacaine Collagen Sponge (CollaRx®) — The bupivacaine sponge contains 70 mg Type I collagen and 50 mg bupivacaine hydrochloride. A total of 3 sponges will be implanted during surgery; one sponge divided between areas in the vault, one sponge divided and placed across the incision in the peritoneum and the final sponge divided and placed between the sheath and skin around the incision.
  Other Names: CollRx Bupivacaine Implant
  Arms: 1
Drug: placebo — The placebo sponge contains 70 mg Type I collagen. A total of 3 sponges will be implanted during surgery; one sponge divided between areas in the vault, one sponge divided and placed across the incision in the peritoneum and the final sponge divided and placed between the sheath and skin around the incision.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the CollaRx Bupivacaine implant is safe and effective in reducing the amount of narcotic pain medication needed to control pain during the first 24 hours after abdominal hysterectomy surgery.

DETAILED DESCRIPTION:
Hysterectomy is the second most common surgery among women in the United States (US). According to the National Center for Health Statistics, there were 617,000 hysterectomies performed in the US in 2004. Effective postoperative pain management after hysterectomy is important in ensuring that surgical subjects have a smooth and successful recovery after their operation. Morphine and other narcotic pain medications are often used to help control pain after hysterectomy, but the large quantities required can lead to fatigue, nausea and vomiting, as well as the inability to walk around much because of drowsiness. Reducing narcotic pain medication use can reduce these negative side effects.

Bupivacaine is a local anesthetic (pain medicine) that has an established safety profile. Collagen is a protein that is found in all mammals. The CollaRx Bupivacaine implant is a thin flat sponge made out of collagen that comes from cow tendons and contains bupivacaine. When inserted into a surgical site, the collagen breaks down and bupivacaine is released at the site but very little is absorbed into the blood stream. The high levels of bupivacaine at the surgical site may result in less pain for several days after surgery.

This study will compare the amount of narcotic pain medication required after surgery in patients who receive the CollaRx Bupivacaine implant, a plain collagen implant or no implant at all.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) > 19 and < 40 kg/m2
* Had planned an elective total abdominal hysterectomy for reasons other than malignancies to be performed according to standard surgical technique using a standard incision and under general anesthesia with the following caveats:

  1. Laparoscopic procedures or supraumbilical or Maylard incisions will not be allowed
  2. A nonlaparoscopic incision for benign non-hysterectomy gynecological procedures (such as myomectomy or adnexal surgery) is acceptable if the surgical indication is not to treat pelvic pain
  3. No concomitant vaginal procedures are allowed. An abdominal urethropexy and an incidental appendectomy will be allowed
* Have a risk classification of I, II or III according to the American Society of Anesthesiologists (ASA)
* Have a negative pregnancy test
* Be free of other physical or mental conditions which may confound assessment of postoperative pain
* Have the ability to read, understand and comply with the study procedures and the use of the pain scales; is capable of operating a patient-controlled analgesia (PCA) device; and is able to communicate meaningfully with the study staff
* Voluntarily sign and date an informed consent form (ICF), prior to the conduct of any study-specific procedures
* Able to fluently speak and understand English and be able to provide meaningful written informed consent for the study

Exclusion Criteria:

* Known hypersensitivity to any active or inactive ingredient of the test articles
* Presence of clinically significant cardiac arrhythmias or atrioventricular (AV) conduction disorders
* Concomitant use of other amide local anesthetics
* Concomitant use of antiarrhythmics
* Concomitant use of propanolol
* Concomitant use of strong/moderate CYP3A4 inhibitors or inducers
* Has used aspirin or aspirin-containing products within 7 days of surgery.
* Previous major surgery in the last 3 months
* Requires any additional surgical procedures during the same hospitalization (except as noted)
* Received neuraxial (spinal or epidural) opioid analgesics either prior to or during surgery
* Received local anesthetic infiltration of the surgical wound prior to, during or immediately after closure
* Is scheduled to receive local anesthetics via an indwelling catheter after surgery
* Underwent additional procedures during surgery, which may increase the visceral pain
* Has known or suspected history of alcohol or drug abuse or misuse or evidence for tolerance or physical dependency on opioids analgesics or sedative-hypnotic medications
* Uses opioids or tramadol daily for > 7 days prior to test article administration
* Has impaired liver function
* Has any clinically significant unstable condition that could compromise the patient's welfare
* Is at risk for infection or slow wound healing
* Has a chronic painful condition that might confound the assessment of pain associated with the sugery
* Has taken pain medication that could confound the analgesic responses the day of surgery
* Has been treated within 2 weeks of surgery with agents that could affect the analgesic response
* Has been treated with monoamine oxidase inhibitors (MAOIs) or MAOIs have been stopped fewer than 10 days prior to surgery
* Has been treated with corticosteroids or whose treatment with these has been stopped < 7 days prior surgery (inhaled corticosteroids are acceptable)
* Has participated in a clinical trial in the previous 30 days
* Has been hemodynamically unstable at any point in the previous 4 weeks or becomes hemodynamically unstable during surgery
* Required blood transfusion in the previous month, except as related to uterine bleeding caused by uterine fibroids.
* Has hemoglobin levels < 10 g/dL or < 8 g/dL for patients with an anemia secondary to heavy uterine bleeding caused by uterine fibroids.
* Has platelet count < 100,000/mm
* Unreliable or incapable of complying with the protocol

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-12-27 (Actual); Primary Completion 2008-09-05 (Actual); Study Completion 2008-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, Study Director — Innocoll
Locations (1):
- Forsyth Medical Centre - OB Anesthesia, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine Sponges: A total of three 5 × 5-cm bupivacaine sponges implanted at specified layers in the wound prior to wound closure
  Bupivacaine Collagen Sponge (CollaRx®): The bupivacaine sponge contains 70 mg Type I collagen and 50 mg bupivacaine hydrochloride. A total of 3 sponges will be implanted during surgery; one sponge divided between areas in the vault, one sponge divided and placed across the incision in the peritoneum and the final sponge divided and placed between the sheath and skin around the incision.
- Collagen Sponges: A total of three 5 × 5-cm collagen sponges implanted at specified layers in the wound prior to wound closure
  placebo: The placebo sponge contains 70 mg Type I collagen. A total of 3 sponges will be implanted during surgery; one sponge divided between areas in the vault, one sponge divided and placed across the incision in the peritoneum and the final sponge divided and placed between the sheath and skin around the incision.
- Standard of Care no Implant: The patient will receive the standard of care, but no implant during surgery
Period: Overall Study
Arm/Group | Bupivacaine Sponges | Collagen Sponges | Standard of Care no Implant
Started | 28 | 15 | 11
Completed | 28 | 15 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Sponges | Collagen Sponges | Standard of Care no Implant | Total
Number analyzed (Participants) | 28 | 15 | 11 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (6.87) | 39.7 (7.06) | 42.9 (6.17) | 42.2 (42.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 15 | 11 | 54
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 3 | 17
  White | 21 | 7 | 7 | 35
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Use of Opioid Rescue Analgesia
Description: Total use of opioid rescue analgesia (mg equivalent) -higher score means more analgesia was needed and worse outcome
Time Frame: 0 to 24 hours postoperatively
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | Bupivacaine Sponges | Collagen Sponges | Standard of Care no Implant
Number analyzed (Participants) | 28 | 15 | 11
mg morphine equivalents | 53.65 (32.78) | 66.56 (47.53) | 53.73 (47.71)

2. Secondary Outcome: Total Use of Opioid Rescue Analgesia
Description: Total use of opioid rescue analgesia (mg equivalent) -higher score means more analgesia was needed and worse outcome
Time Frame: 0 to 48 hours postoperatively
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | Bupivacaine Sponges | Collagen Sponges | Standard of Care no Implant
Number analyzed (Participants) | 28 | 15 | 11
mg morphine equivalents | 67.78 (37.195) | 80.87 (51.085) | 66.03 (32.41)

3. Secondary Outcome: Total Use of Opioid Rescue Analgesia
Description: Total use of opioid rescue analgesia (mg equivalent) -higher score means more analgesia was needed and worse outcome
Time Frame: 0 to 72 hours postoperatively
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | Bupivacaine Sponges | Collagen Sponges | Standard of Care no Implant
Number analyzed (Participants) | 28 | 15 | 11
mg morphine equivalents | 78.13 (40.304) | 88.60 (55.84) | 73.28 (36.308)

4. Secondary Outcome: Pain Intensity Rating on a Visual Analog Scale (at Rest)
Description: Pain intensity rating on a Visual Analog Scale (at rest). Lowest score possible is "0" with the highest score possible being "100". Higher number means more pain reported.
Time Frame: At 1, 1.5, 2, 3, 6, 9, 12, 18, 24, 36, 48 and 72 hours post operatively
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Sponges | Collagen Sponges | Standard of Care no Implant
Number analyzed (Participants) | 28 | 15 | 11
score on a scale
  Hour 1.0 | 58.5 (33.59) | 63.0 (30.08) | 66.5 (30.29)
  Hour 1.5 | 60.1 (29.88) | 61.3 (31.48) | 61.3 (32.68)
  Hour 2.0 | 54.2 (23.92) | 50.3 (28.93) | 61.9 (28.39)
  Hour 3.0 | 47.0 (28.27) | 46.2 (31.80) | 46.4 (31.57)
  Hour 6.0 | 38.5 (24.47) | 43.3 (32.49) | 34.7 (27.17)
  Hour 9.0 | 36.2 (25.22) | 39.9 (31.49) | 44.0 (31.07)
  Hour 12 | 36.1 (24.79) | 32.4 (26.40) | 38.4 (32.21)
  Hour 18 | 41.6 (22.45) | 29.8 (29.78) | 24.0 (24.64)
  Hour 24 | 33.3 (24.71) | 32.0 (31.07) | 41.7 (39.29)
  Hour 36 | 32.6 (23.27) | 18.7 (18.40) | 41.8 (39.03)
  Hour 48 | 26.4 (20.41) | 26.7 (26.91) | 22.2 (29.41)
  Hour 72 | 18.6 (16.03) | 14.7 (17.43) | 27.7 (29.57)

5. Secondary Outcome: Time to First Use of Opioid Rescue Analgesia
Description: Time to first use of opioid rescue analgesia - lower number means worse outcome
Time Frame: Actual time assessed during post operative period
Population: Intent-to-Treat Population
Measure: Median (95% Confidence Interval); unit: Time (Hours)
Arm/Group | Bupivacaine Sponges | Collagen Sponges | Standard of Care no Implant
Number analyzed (Participants) | 28 | 15 | 11
Time (Hours) | 0.9 [0.8 to 1.3] | 0.9 [0.6 to 1.1] | 0.4 [0.2 to 1.0]

6. Secondary Outcome: Pain Intensity Rating on a Visual Analog Scale (After Cough)
Description: Pain intensity rating on a Visual Analog Scale (after cough). Lowest score possible is "0" with the highest score possible being "100". Higher number means more pain reported.
Time Frame: At 1, 1.5, 2, 3, 6, 9, 12, 18, 24, 36, 48 and 72 hours post operatively
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Sponges | Collagen Sponges | Standard of Care no Implant
Number analyzed (Participants) | 28 | 15 | 11
score on a scale
  Hour 1.0 | 68.2 (32.96) | 73.8 (33.55) | 72.6 (31.01)
  Hour 1.5 | 68.2 (29.49) | 67.3 (34.05) | 73.8 (27.44)
  Hour 2.0 | 66.0 (24.96) | 61.3 (32.17) | 72.9 (26.08)
  Hour 3.0 | 53.9 (29.02) | 58.0 (32.82) | 59.0 (30.29)
  Hour 6.0 | 48.3 (27.73) | 64.7 (31.63) | 53.2 (29.86)
  Hour 9.0 | 52.8 (27.69) | 49.8 (29.12) | 63.1 (22.64)
  Hour 12 | 52.5 (24.56) | 49.1 (26.22) | 55.0 (27.19)
  Hour 18 | 55.8 (25.40) | 46.7 (28.79) | 45.3 (28.08)
  Hour 24 | 46.8 (26.65) | 52.0 (32.14) | 59.1 (30.58)
  Hour 36 | 51.2 (28.06) | 32.0 (23.81) | 58.2 (34.69)
  Hour 48 | 40.7 (29.30) | 46.8 (27.24) | 38.0 (27.80)
  Hour 72 | 28.0 (25.97) | 28.6 (27.94) | 40.1 (30.85)

7. Secondary Outcome: Pain Intensity Rating on a 4-point Likert Scale (at Rest)
Description: For the 4-point categorical scale assessment, patients measured their pain intensity at rest using a numerical scale where: 0 = "none," 1 = "mild," 2 = "moderate" and 3 = "severe."
Time Frame: At 1, 1.5, 2, 3, 6, 9, 12, 18, 24, 36, 48 and 72 hours post operatively
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Sponges | Collagen Sponges | Standard of Care no Implant
Number analyzed (Participants) | 28 | 15 | 11
score on a scale
  Hour 0.5 | 1.8 (1.00) | 2.0 (1.00) | 2.2 (1.03)
  Hour 1.0 | 2.0 (0.95) | 2.2 (0.69) | 2.2 (0.79)
  Hour 1.5 | 2.0 (0.79) | 2.0 (0.88) | 2.1 (0.83)
  Hour 2.0 | 2.0 (0.62) | 1.7 (0.70) | 2.0 (0.77)
  Hour 3.0 | 1.7 (0.71) | 1.6 (0.74) | 1.9 (0.88)
  Hour 6.0 | 1.5 (0.64) | 1.3 (0.96) | 1.6 (0.52)
  Hour 9.0 | 1.4 (0.63) | 1.5 (0.83) | 1.8 (0.83)
  Hour 12 | 1.4 (0.75) | 1.1 (0.64) | 1.7 (0.76)
  Hour 18 | 1.5 (0.51) | 1.1 (0.74) | 1.4 (0.79)
  Hour 24 | 1.3 (0.75) | 1.1 (0.70) | 1.5 (0.82)
  Hour 36 | 1.3 (0.82) | 0.8 (0.43) | 1.4 (0.52)
  Hour 48 | 1.1 (0.63) | 0.9 (0.70) | 0.9 (0.83)
  Hour 72 | 0.9 (0.69) | 0.6 (0.63) | 1.1 (0.70)

8. Secondary Outcome: Pain Intensity Rating on a 4-point Likert Scale (After Cough)
Description: For the 4-point categorical scale assessment, patients measured their pain intensity after aggravated movement (cough) using a numerical scale where: 0 = "none," 1 = "mild," 2 = "moderate" and 3 = "severe."
Time Frame: At 1, 1.5, 2, 3, 6, 9, 12, 18, 24, 36, 48 and 72 hours post operatively
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Sponges | Collagen Sponges | Standard of Care no Implant
Number analyzed (Participants) | 28 | 15 | 11
score on a scale
  Hour 0.5 | 2.1 (1.02) | 2.2 (0.83) | 2.4 (0.84)
  Hour 1.0 | 2.2 (0.95) | 2.5 (0.78) | 2.4 (0.84)
  Hour 1.5 | 2.2 (0.83) | 2.2 (0.80) | 2.5 (0.69)
  Hour 2.0 | 2.2 (0.66) | 2.0 (0.93) | 2.3 (0.79)
  Hour 3.0 | 2.1 (0.80) | 2.1 (0.88) | 2.2 (0.79)
  Hour 6.0 | 1.8 (0.75) | 2.1 (0.74) | 2.1 (0.57)
  Hour 9.0 | 1.9 (0.74) | 2.1 (0.80) | 2.2 (0.67)
  Hour 12 | 1.9 (0.91) | 1.8 (0.69) | 2.0 (0.58)
  Hour 18 | 1.8 (0.73) | 1.9 (0.74) | 1.7 (0.76)
  Hour 24 | 1.7 (0.76) | 1.8 (0.77) | 1.9 (0.57)
  Hour 36 | 1.8 (0.87) | 1.4 (0.76) | 1.9 (0.74)
  Hour 48 | 1.5 (0.84) | 1.5 (0.92) | 1.5 (0.69)
  Hour 72 | 1.3 (0.68) | 1.3 (0.49) | 1.3 (0.79)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Bupivacaine Sponges | Collagen Sponges | Standard of Care no Implant
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/15 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/28 | 0/15 | 1/11
Other Adverse Events (participants affected / at risk) | 21/28 | 12/15 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine Sponges (N=28) | Collagen Sponges (N=15) | Standard of Care no Implant (N=11)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine Sponges (N=28) | Collagen Sponges (N=15) | Standard of Care no Implant (N=11)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 13 (13) | 10 (10) | 5 (5)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No